CLINICAL TRIAL: NCT06849973
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2/ Phase 3 Study of NA-921 (Bionetide) for the Treatment of Girls and Women with Rett Syndrome
Brief Title: To Study the Efficacy & Safety of Oral NA-921 (Bionetide) in Girls and Women with Rett Syndrome
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biomed Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2024-R01
Record Dates: First submitted 2025-02-24; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome; Mental Retardation, X-Linked; Genetic Diseases, X-Linked
MeSH Terms: conditions — Rett Syndrome; X-Linked Intellectual Disability; Genetic Diseases, X-Linked

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Drug - NA-921 (Bionetide) (Experimental): NA-921 (Bionetide) solution of 20-40 mL based on the subject's weight at Basel
  Interventions: Drug: Drug: Bionetide
- Placebo Comparator: Placebo (Placebo Comparator): Bionetide placebo solution of 20-40 mL based on the subject's weight at Baseline, administered twice daily by mouth or gastrostomy tube (G-tube)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Drug: Bionetide — NA-921 (Bionetide) solution administered based on the subject's weight at Baseline, twice daily for 12 weeks
  Other Names: NA-921
  Arms: Experimental: Drug - NA-921 (Bionetide)
Drug: Placebo — NA-921 (Bionetide) placebo solution administered based on the subject's weight at Baseline, twice daily for 12 weeks
  Other Names: NA-921 placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
To study the efficacy & safety of oral Bionetide versus placebo in girls and women with Rett syndrome

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Phase 2/3 Study of NA-921 (Bionetide) for the Treatment of Girls and Women with Rett Syndrome

Primary Objective • To investigate the efficacy and safety of treatment with oral NA-921 (Bionetide) versus placebo in girls and women with Rett syndrome

Key Secondary Objective • To investigate the efficacy of treatment with oral NA-921 (Bionetide) versus placebo on ability to communicate in girls and women with Rett syndrome

Co-Primary Endpoints

* Rett Syndrome Behavior Questionnaire (RSBQ) total score - Change from Baseline to Week 12
* Clinical Global Impression-Improvement (CGI-I) Score at Week 12

Key Secondary Endpoint

Change from Baseline to Week 12 in:

• Communication and Symbolic Behavior Scales Developmental Profile™ Infant-Toddler Checklist- Social Composite Score (CSBS-DP-IT Social)

ELIGIBILITY:
INCLUSION CRITERIA:

* Female subjects 5 to 20 years of age, inclusive, at Screening
* Body weight ≥12 kg at Screening
* Can swallow the study medication provided as a liquid solution or can take it by gastrostomy tube
* Has classic/typical Rett syndrome (RTT)
* Has a documented disease-causing mutation in the MECP2 gene
* Has a stable pattern of seizures, or has had no seizures, within 8 weeks of Screening
* Subjects of childbearing potential must abstain from sexual activity for the duration of the study and for at least 30 days thereafter or must agree to use acceptable methods of contraception. Subject must not be pregnant or breastfeeding.
* The subject's caregiver is English-speaking and has sufficient language skills to complete the caregiver assessments
* Subject and caregiver(s) must reside at a location to which study drug can be delivered and have been at their present residence for at least 3 months prior to Screening

EXCLUSION CRITERIA :

* Has been treated with insulin within 12 weeks of Baseline
* Has current clinically significant cardiovascular, endocrine (such as hypo- or hyperthyroidism, Type 1 diabetes mellitus, or uncontrolled Type 2 diabetes mellitus), renal, hepatic, respiratory or gastrointestinal disease (such as celiac disease or inflammatory bowel disease) or has major surgery planned during the study
* Has a history of, or current, cerebrovascular disease or brain trauma
* Has significant, uncorrected visual or uncorrected hearing impairment
* Has a history of, or current, malignancy
* Has a known history or symptoms of long QT syndrome

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all pre-specified entry criteria).

Ages: 5 Years to 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female
Enrollment: 187 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-01-28 (Actual)

PRIMARY OUTCOMES:
Rett Syndrome Behavior Questionnaire (RSBQ) Total Score - Change From Baseline to Week 12 | Baseline and Week 12
  The RSBQ is a 45-item caregiver-completed rating scale that includes 45 items, 39 of them grouped into 8 subscales, whose ratings reflect the severity and frequency of symptoms. Items are rated as 0 (not true), 1 (somewhat or sometimes true), or 2 (very true). The 8 subscales are general mood, breathing problems, hand behavior, face movements, body rocking/expressionless face, night-time behaviors, fear/anxiety, and walking/standing. Scores for item 31 are reversed in the calculation of the total score. The total score ranges from 0 to 90 and is calculated as the sum of the item scores. Higher scores mean worse behavior.
Clinical Global Impression-Improvement (CGI-I) Score at Week 12 | 12 Weeks Treatment Duration
  To rate how much the subject's illness has improved or worsened relative to a baseline state, a 7-point scale is used from 1=very much improved, 2=much improved, 3=minimally improved, 4=no change, 5=minimally worse, 6=much worse, 7=very much worse.

SECONDARY OUTCOMES:
Change From Baseline to Week 12 in Communication and Symbolic Behavior Scales Developmental Profile™ Infant-Toddler Checklist - Social Composite Score (CSBS-DP-IT Social) | 12 Weeks Treatment Duration
  Standardized screening scale for assessing communication and pre-linguistic skills in young children 12-24 months and can be used with older children with developmental delay. The CSBS-DP includes a suite of three separate measures: The Infant-Toddler Checklist, a follow-up Caregiver Questionnaire and a Behavior Sample. In this study only the Infant-Toddler (CSBS-DP-IT) Checklist was used. The CSBS-DP-IT Checklist is a 24-item rating scale and each item is scored using a three-level rating of frequency: "not yet", "sometimes" and "often". The CSBS-DP-IT Social Composite score the range was 0 to 26 and a higher score represented a worse outcome. Three composite scores can be calculated: 1) Social Composite; 2) Speech Composite; 3) Symbolic Composite.
Change From Baseline to Week 12 in Rett Syndrome Clinician Rating of Ability to Communicate Choices (RTT-COMC) | 12 Weeks Treatment Duration
  Clinical assessment of the subject's ability to communicate their choices or preferences, which can include the use of nonverbal means such as eye contact or gestures. The assessment is made on an 8-point Likert scale (0-7) with 0 denoting normal functioning and 7 the most severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Lloyd L. Tran, PhD, Study Director — Biomed Industries, Inc.; David Nguyen, PhD, Study Director — Biomed Industries, Inc.
Locations (16):
- United States (12):
  - Biomed Testing Facility # BIO-04-92093, La Jolla, California
  - Biomed Testing Facility # BIO-03-90095, Los Angeles, California
  - Biomed Testing Facility # BIO-02-95817, Sacramento, California
  - Biomed Testing Facility # BIO-01-94104, San Francisco, California
  - Biomed Testing Facility #BIO-05-80042, Aurora, Colorado
  - Biomed Testing Facility #BIO-06-60612, Chicago, Illinois
  - Maryland Locations Biomed Testing Facility #BIO-7-21205, Baltimore, Maryland
  - Biomed Testing Facility #BIO-8-02115, Boston, Massachusetts
  - Biomed Testing Facility #BIO-9-10467, The Bronx, New York
  - Biomed Testing Facility #BIO-10-44195, Cleveland, Ohio
  - Biomed Testing Facility #BIO-11-77030, Houston, Texas
  - Biomed Testing Facility #BIO-12-98105, Seattle, Washington
- Australia (4):
  - Biomed Research Unit-BIO-16-NSW, Camperdown, New South Wales
  - Biomed Research Unit-BIO-15, Sydney, New South Wales
  - Biomed Research Unit-BIO-13-VIC-3084 Heidelberg West, Victoria, Australia, 3084, Heidelberg West, Victoria
  - Biomed Research Unit- BIO-14-VIC 3010, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
We will decide whether to share IPD at a later date